CLINICAL TRIAL: NCT00425269
Title: Evaluation of a Lifestyle Intervention to Prevent Type 2 Diabetes/Metabolic Syndrome Among Pakistani Immigrants - Focusing on Changes in Diet and Physical Activity
Brief Title: Lifestyle Intervention for Pakistani Women in Oslo
Acronym: InnvaDiab
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oslo (Other)
Collaborators: European Commission (Other); The Research Council of Norway (Other)
Responsible Party: Principal Investigator, Gerd Holmboe-Ottesen, PhD, University of Oslo
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: NFR 166998/166977; EU-DEPLAN 2004310
Record Dates: First submitted 2007-01-19; First posted 2007-01-22 (Estimated); Results first posted 2014-07-21 (Estimated); Last update posted 2014-07-21 (Estimated); Status verified 2014-04

CONDITIONS: Metabolic Syndrome; Type 2 Diabetes
Keywords: lifestyle intervention; Type 2 Diabetes; Metabolic syndrome; Pakistani women; dietary change; Physical activity; Norway
MeSH Terms: conditions — Metabolic Syndrome; Diabetes Mellitus, Type 2; Motor Activity | interventions — Diet; Exercise

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Experimental): The intervention group was divided into nine subgroups of ten to twelve women who were offered six educational sessions, each lasting 2 h, during a 7 +- 1-month period. The main focus was on the physiological importance of blood glucose and its regulation by diet and physical activity, and on knowledge about the Pakistani lifestyle in Pakistan and Norway
  Interventions: Behavioral: lifestyle intervention (diet and physical activity)
- Control (No Intervention): One lesson recieved after post-test

INTERVENTIONS:
Behavioral: lifestyle intervention (diet and physical activity) — The intervention will include a combination of individual counselling group sessions. The intervention groups will be divided into subgroups of 10-12 subjects. Each group will have 10 group sessions on diet/lifestyle in the 6 months the intervention period lasts, and will additionally have the possibility to join a culturally adapted exercise program of low intensity twice a week.
  Arms: Intervention

SUMMARY:
Immigrants from South Asia in Norway have a high prevalence of type 2 diabetes and conditions related to the metabolic syndrome. It has been documented that these conditions may be prevented by changes in lifestyle. No previous intervention studies on immigrants with focus on diet and physical activity have been carried out in Norway. This project concerns a randomized controlled trial with intervention to change diet and physical activity in 200 high risk female Pakistani immigrants living in Oslo. The intervention will be evaluated both in terms of outcome and process.

DETAILED DESCRIPTION:
Objectives:

1. To evaluate the health effects of systematic dietary education and counselling and physical training in a group of Pakistani women with high risk of type 2 diabetes.
2. To evaluate the intervention process in order to identify the most effective methods of intervention in regard to diet and physical activity for immigrant women of Pakistani origin.

Background: Immigrants from South Asia have a high prevalence of type 2 diabetes, which may be prevented by intensive on physical activity and diet. This application concerns intervention with diet and physical activity in female (ongoing study) and male (extended study) Pakistani immigrants living in Oslo to reduce their risk for these diseases.

Intervention design: The subjects will be 200 women randomized into an intervention group and a control group (100 in each). The women are being recruited from a township in Oslo with a high proportion of immigrants by using a network approach. Inclusion criteria is based on a risk score developed by Ramachandran et al for Asian Indians, entailing age, Body Mass Index, waist circumference, family history of diabetes and sedentary physical activity.

The intervention will include a combination of individual counselling and group sessions. The intervention group will be divided into subgroups of 10-12 subjects. Each subgroup will have 10 group sessions on diet/lifestyle in the 6 months the intervention period lasts, and will additionally have the possibility to join a cultural adapted exercise program of low intensity twice a week. This includes indoor activities (exercise with music) and outdoor activities (walking groups).

Evaluation: The main end point of the intervention will be the fasting and 2-h plasma glucose value after an oral glucose tolerance test (OGTT). This will be measured at baseline and after 6 months of intervention.

Secondary end-points will be Serum lipid profile (e.g. triglycerides, High-Density Lipoprotein-cholesterol) ; HbA1c ; C-peptide ; serum insulin; serum albumin; body weight; waist and hip circumference; maximum heart rate on treadmill test; self-reported level of intensity, duration and frequency of physical activity; self-reported level of "Stages of change" in regard to motivation and behavioural change; self- reported subjective health complaints; self-reported coping strategies; self-reported sleeping habits.

Dietary information will be collected by 2 x 48 hours dietary recalls. The intake of energy and nutrients will be calculated from the recalls, as well as the intake of food groups.The diet will also be evaluated by a culturally adapted food frequency questionnaire including 20 food groups (with portion sizes). In addition, the use of cooking oils will be registered by questions about the type and quantity oil used per time unit in the household. Additionally, information on knowledge and perceptions on diet and health before and after the intervention will be registered.

Physical activity will be registered using an advanced continuous body monitor, SenseWear Armband yielding information on total energy expenditure, level of intensity, duration and frequency of physical activity, duration of lying down, duration of sleeping, and sleeping quality.

The completion of the questionnaires will take the form of an interview by Urdu speaking staff.

ELIGIBILITY:
Inclusion Criteria:

* Risk score developed by Ramachandran et al for Asian Indians:

  * BMI, waist circumference, family history of diabetes and sedentary physical activity

Exclusion Criteria:

* Type 1 diabetes.
* Positive auto antibodies.
* Diagnosis of type 2 diabetes more than 6 months.
* Medication for type 2 diabetes.
* Pregnancy at intervention start.
* Suffering from heart attack or stroke the last 3 months.
* Already participating in organised physical exercise.

Min Age: 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 198 (Actual)
Dates: Start 2006-04; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gerd Holmboe-Ottesen, Dr. Philos., Principal Investigator — University of Oslo
Locations (1):
- Primary Health Care Health Center, Oslo, Holmlia, Oslo, Norway

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A multi-recruitment strategy included visits to mosques and other formal and informal gatherings in the local community, as well as word of mouth. Interested women came to an appointment at the local mother and baby health care centre where the intervention took place. An Urdu-speaking research assistant was in charge of the recruitment
Groups:
- Intervention: Intervention Group (n 101) The women in the intervention group was divided into nine subgroups of 10-12 women. Each subgroup had six group sessions, lasting 2 h each, during the 7 ± 1 month of the intervention.
  The group sessions were focused on the importance of diet and physical activity for blood glucose regulation. They aimed at helping the women to incorporate the knowledge acquired into their everyday lives, and to help the women obtaining positive expectancies for lifestyle changes. Culturally adapted materials were used and discussions were encouraged. All the teaching was translated into Punjabi, the preferred language of the participants.
- Control: Control Group (n 97) The women in the control group received one group teaching with the main points after the follow-up tests.
Period: Overall Study
Arm/Group | Intervention | Control
Started | 101 | 97
Completed | 82 | 77
Not Completed | 19 | 20
Not completed — Pregnancy | 5 | 7
Not completed — Lost to Follow-up | 9 | 9
Not completed — moved or medical reason | 5 | 4

BASELINE CHARACTERISTICS:
Population: Women, aged 18-65 years, more than 50 percent rated their command of the Norwegian language as poor, and mean number of years of education was 9.
Groups:
- Total: Total of all reporting groups
Arm/Group | Intervention | Control | Total
Number analyzed (Participants) | 101 | 97 | 198
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 101 | 97 | 198
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 101 | 97 | 198
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Norway | 101 | 97 | 198
Years of residence in Norway [Mean (Standard Deviation); unit: years] | 18 (7.9) | 19 (7.6) | 19 (7.8)
Years of education [Mean (Standard Deviation); unit: years] | 9 (4.7) | 9 (4.3) | 9 (4.5)
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 29.4 (5.6) | 29.8 (5.5) | 29.6 (5.6)

OUTCOME MEASURES:

1. Primary Outcome: The Fasting Plasma Glucose Value, Baseline
Time Frame: baseline
Measure: Mean (95% Confidence Interval); unit: mmol/L
Groups:
- Control: Control Group (n 97) The women in the control group recieved one group teaching with the main points after the follow-up tests.
Arm/Group | Intervention | Control
Number analyzed (Participants) | 101 | 97
mmol/L | 5.55 [5.37 to 5.72] | 5.53 [5.37 to 5.69]

2. Primary Outcome: Plasma Glucose 2 h After Oral Glucose Tolerance Test, Baseline
Time Frame: baseline
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Intervention | Control
Number analyzed (Participants) | 101 | 97
mmol/L | 8.52 [8.03 to 9.02] | 8.41 [7.86 to 8.96]

3. Secondary Outcome: HbA1c, Baseline
Time Frame: baseline
Measure: Mean (95% Confidence Interval); unit: percent of Hb
Arm/Group | Intervention | Control
Number analyzed (Participants) | 101 | 97
percent of Hb | 5.4 [5.3 to 5.5] | 5.4 [5.3 to 5.5]

4. Secondary Outcome: C-peptide, 0-h, Baseline
Time Frame: baseline
Measure: Mean (95% Confidence Interval); unit: pmol/L
Arm/Group | Intervention | Control
Number analyzed (Participants) | 101 | 97
pmol/L | 855.0 [787.2 to 922.8] | 839.9 [769.3 to 910.5]

5. Secondary Outcome: C-peptid, 2-h, Baseline
Time Frame: baseline
Measure: Mean (95% Confidence Interval); unit: pmol/L
Arm/Group | Intervention | Control
Number analyzed (Participants) | 101 | 97
pmol/L | 3851.5 [3508.1 to 4194.9] | 3628.9 [3258.2 to 3999.5]

6. Secondary Outcome: Insulin, 0-h, Baseline
Time Frame: baseline
Measure: Mean (95% Confidence Interval); unit: pmol/L
Arm/Group | Intervention | Control
Number analyzed (Participants) | 101 | 97
pmol/L | 127.6 [113.6 to 141.7] | 116.3 [103.9 to 128.6]

7. Secondary Outcome: Insulin, 2-h, Baseline
Time Frame: baseline
Measure: Mean (95% Confidence Interval); unit: pmol/L
Arm/Group | Intervention | Control
Number analyzed (Participants) | 101 | 97
pmol/L | 931.1 [715.2 to 1146.7] | 839.5 [593.6 to 1085.4]

8. Secondary Outcome: High-Density Lipoprotein Cholesterol, Baseline
Time Frame: baseline
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Intervention | Control
Number analyzed (Participants) | 101 | 97
mmol/L | 1.26 [1.20 to 1.33] | 1.25 [1.19 to 1.32]

9. Secondary Outcome: Triglycerides, Baseline
Time Frame: baseline
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Intervention | Control
Number analyzed (Participants) | 101 | 97
mmol/L | 1.4 [1.2 to 1.5] | 1.4 [1.3 to 1.5]

10. Secondary Outcome: Systolic Blood Pressure, Baseline
Time Frame: baseline
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Intervention | Control
Number analyzed (Participants) | 101 | 97
mmHg | 115.6 [111.7 to 119.6] | 118.7 [115.5 to 122.0]

11. Secondary Outcome: Diastolic Blood Pressure, Baseline
Time Frame: baseline
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Intervention | Control
Number analyzed (Participants) | 101 | 97
mmHg | 80.0 [77.8 to 82.4] | 80.8 [78.9 to 82.7]

12. Secondary Outcome: Waist Circumference, Baseline
Time Frame: baseline
Measure: Mean (95% Confidence Interval); unit: cm
Arm/Group | Intervention | Control
Number analyzed (Participants) | 101 | 97
cm | 95.3 [92.4 to 98.1] | 96.2 [93.9 to 98.5]

13. Secondary Outcome: Body Mass Index, Baseline
Time Frame: baseline
Measure: Mean (95% Confidence Interval); unit: kg/m^2
Arm/Group | Intervention | Control
Number analyzed (Participants) | 101 | 97
kg/m^2 | 29.39 [28.3 to 30.6] | 29.73 [28.6 to 30.9]

14. Secondary Outcome: Intake of Vegetables, Fruit and Fruit Juice, Baseline
Time Frame: baseline
Measure: Mean (Inter-Quartile Range); unit: gram per day
Arm/Group | Intervention | Control
Number analyzed (Participants) | 101 | 97
gram per day | 328.9 [161 to 450] | 306.3 [193 to 375]

15. Secondary Outcome: Intake of Soft Drinks With Added Sugar, Baseline
Time Frame: baseline
Measure: Mean (Inter-Quartile Range); unit: dL/week
Arm/Group | Intervention | Control
Number analyzed (Participants) | 101 | 97
dL/week | 5.0 [0.0 to 5.8] | 4.4 [0.0 to 5.8]

16. Secondary Outcome: Intake of Red Meat, Baseline
Time Frame: baseline
Measure: Mean (Inter-Quartile Range); unit: portions/week
Arm/Group | Intervention | Control
Number analyzed (Participants) | 101 | 97
portions/week | 2.1 [1.0 to 2.5] | 2.0 [1.0 to 2.5]

17. Secondary Outcome: Intake of Poultry, Baseline
Time Frame: baseline
Measure: Mean (Inter-Quartile Range); unit: portions/week
Arm/Group | Intervention | Control
Number analyzed (Participants) | 101 | 97
portions/week | 2.1 [1.0 to 3.0] | 2.1 [1.0 to 2.5]

18. Secondary Outcome: Intake of Fish, Baseline
Time Frame: baseline
Measure: Mean (Inter-Quartile Range); unit: portions/week
Arm/Group | Intervention | Control
Number analyzed (Participants) | 101 | 97
portions/week | 0.97 [0.38 to 1.3] | 0.77 [0.0 to 1.0]

19. Primary Outcome: The Fasting Plasma Glucose, Post-test
Time Frame: post-test
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Intervention | Control
Number analyzed (Participants) | 82 | 77
mmol/L | 5.39 [5.24 to 5.54] | 5.66 [5.36 to 5.95]

20. Primary Outcome: Plasma Glucose, 2-h, Post-test
Time Frame: post-test
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Intervention | Control
Number analyzed (Participants) | 82 | 77
mmol/L | 8.00 [7.52 to 8.48] | 8.20 [7.58 to 8.80]

21. Secondary Outcome: HbA1C, Post-test
Time Frame: post-test, after completion of all six group sessions
Measure: Mean (95% Confidence Interval); unit: percent of Hb
Arm/Group | Intervention | Control
Number analyzed (Participants) | 82 | 77
percent of Hb | 5.4 [5.3 to 5.5] | 5.5 [5.3 to 5.6]

22. Secondary Outcome: C-peptid, 0-h, Post-test
Time Frame: post-test, after completion of all six group sessions
Measure: Mean (95% Confidence Interval); unit: pmol/L
Arm/Group | Intervention | Control
Number analyzed (Participants) | 82 | 77
pmol/L | 878.5 [809.0 to 948.1] | 914.6 [837.8 to 991.5]

23. Secondary Outcome: C-peptid, 2-h, Post-test
Time Frame: post-test, after completion of all six group sessions
Measure: Mean (95% Confidence Interval); unit: pmol/L
Arm/Group | Intervention | Control
Number analyzed (Participants) | 82 | 77
pmol/L | 3618.1 [3297.8 to 3938.3] | 3439.9 [3096.4 to 3783.4]

24. Secondary Outcome: Insulin, 0-h, Post-test
Time Frame: post-test, after completion of all six group sessions
Measure: Mean (95% Confidence Interval); unit: pmol/L
Arm/Group | Intervention | Control
Number analyzed (Participants) | 82 | 77
pmol/L | 121.8 [110.6 to 133.1] | 123.3 [112.1 to 134.5]

25. Secondary Outcome: Insulin, 2-h, Post-test
Time Frame: post-test, after completion of all six group sessions
Measure: Mean (95% Confidence Interval); unit: pmol/L
Arm/Group | Intervention | Control
Number analyzed (Participants) | 82 | 77
pmol/L | 861.8 [660.8 to 1062.8] | 786.1 [615.2 to 957.1]

26. Secondary Outcome: High-Density Lipoprotein Cholesterol, Post-test
Time Frame: post-test, after completion of all six group sessions
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Intervention | Control
Number analyzed (Participants) | 82 | 77
mmol/L | 1.24 [1.17 to 1.30] | 1.20 [1.14 to 1.26]

27. Secondary Outcome: Triglycerides, Post-test
Time Frame: post-test, after completion of all six group sessions
Measure: Mean (95% Confidence Interval); unit: mmol/L
Arm/Group | Intervention | Control
Number analyzed (Participants) | 82 | 77
mmol/L | 1.3 [1.2 to 1.5] | 1.5 [1.3 to 1.6]

28. Secondary Outcome: Systolic Blood Pressure, Post-test
Time Frame: post-test, after completion of all six group sessions
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Intervention | Control
Number analyzed (Participants) | 82 | 77
mmHg | 114.4 [111.0 to 117.7] | 117.1 [114.0 to 120.2]

29. Secondary Outcome: Diastolic Blood Pressure, Post-test
Time Frame: post-test, after completion of all six group sessions
Measure: Mean (95% Confidence Interval); unit: mmHg
Arm/Group | Intervention | Control
Number analyzed (Participants) | 82 | 77
mmHg | 78.6 [76.4 to 80.8] | 80.1 [77.9 to 82.2]

30. Secondary Outcome: Waist Circumference
Time Frame: post-test, after completion of all six group sessions
Measure: Mean (95% Confidence Interval); unit: cm
Arm/Group | Intervention | Control
Number analyzed (Participants) | 82 | 77
cm | 95.1 [92.4 to 97.9] | 96.8 [94.5 to 99.1]

31. Secondary Outcome: Body Mass Index, Post-test
Time Frame: post-test, after completion of all six group sessions
Measure: Mean (95% Confidence Interval); unit: kg/m^2
Arm/Group | Intervention | Control
Number analyzed (Participants) | 82 | 77
kg/m^2 | 29.11 [28.0 to 30.3] | 29.65 [28.5 to 30.8]

32. Secondary Outcome: Intake of Vegetables, Fruit and Fruit Juice, Post-test
Time Frame: post-test, after completion of all six group sessions
Measure: Mean (Inter-Quartile Range); unit: grams per day
Arm/Group | Intervention | Control
Number analyzed (Participants) | 82 | 77
grams per day | 375.4 [193 to 493] | 328.3 [193 to 450]

33. Secondary Outcome: Intake of Soft Drinks With Added Sugar, Post-test
Time Frame: post-test, after completion of all six group sessions
Measure: Mean (Inter-Quartile Range); unit: dl/week
Arm/Group | Intervention | Control
Number analyzed (Participants) | 82 | 77
dl/week | 2.5 [0.0 to 5.8] | 5.1 [0.0 to 5.8]

34. Secondary Outcome: Intake of Red Meat, Post-test
Time Frame: post-test, after completion of all six group sessions
Measure: Mean (Inter-Quartile Range); unit: portions/week
Arm/Group | Intervention | Control
Number analyzed (Participants) | 82 | 77
portions/week | 1.6 [1.0 to 2.0] | 2.0 [1.0 to 2.5]

35. Secondary Outcome: Intake of Poultry, Post-test
Time Frame: post-test, after completion of all six group sessions
Measure: Mean (Inter-Quartile Range); unit: portions/week
Arm/Group | Intervention | Control
Number analyzed (Participants) | 82 | 77
portions/week | 1.9 [1.0 to 2.5] | 1.8 [1.0 to 2.5]

36. Secondary Outcome: Intake of Fish, Post Test
Time Frame: post-test, after completion of all six group sessions
Measure: Mean (Inter-Quartile Range); unit: portions/week
Arm/Group | Intervention | Control
Number analyzed (Participants) | 82 | 77
portions/week | 1.13 [0.5 to 1.5] | 1.11 [0.0 to 2.0]

ADVERSE EVENTS:
Description: serious and/or other [non-serious] adverse events were not collected/assessed
Arm/Group | Intervention | Control
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes